CLINICAL TRIAL: NCT06681831
Title: Feasibility, Safety, and Efficacy of Robotic Single-Port Hysterectomy (R-SPH) Using the Da Vinci SP System in Low-Risk Endometrial Cancer: a Pilot Study
Brief Title: Single-Port Hysterectomy (R-SPH) Using the Da Vinci SP System in Low-Risk Endometrial Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Corrado Giacomo, Principal investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 864/16
Record Dates: First submitted 2024-11-04; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Endometrial Cancer
Keywords: davinci sp; endometrial cancer; robotic surgery
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: DaVinci SP — robotic single-port hysterectomy (R-SPH) with DaVinci SP
  Other Names: robotic singleport surgery

SUMMARY:
Patients with clinically confirmed endometrioid endometrial cancer at FIGO stage IA-IB were eligible for robotic single-port hysterectomy (R-SPH). Criteria included: well or moderately differentiated tumor grade (G1 or G2), sufficient vaginal access, uterine size under 12 weeks' gestation, adequate bone marrow, kidney, liver, and heart function, and an ECOG performance status of 2 or below. Exclusions applied to patients with significant cardiopulmonary disease, previous pelvic or abdominal radiation, or severe hip disease affecting positioning. Prior abdominal surgeries did not exclude patients from robotic surgery. Surgeries were performed using the Vinci Single-Site® system by a specialized team. Clinical data collected included age, BMI, FIGO stage, tumor grade, surgical margin status, and hospital stay duration. Operation times were divided into docking, console (surgical), and total operation times. Intraoperative assessments included complications, blood loss, hemoglobin changes, and transfusions if hemoglobin was ≤7 g/L. Postoperative complications were evaluated short- and long-term, including surgical, cardiac, and respiratory events.

DETAILED DESCRIPTION:
Patients with clinically confirmed endometrioid endometrial cancer, International Federation of Gynaecology and Obstetrics stage IA-IB were eligible for R-SPH. Other eligibility criteria included: tumor grades well (G1) or moderately differentiated (G2) at biopsy; adequate vaginal access and uterine size < 12 weeks gestation; adequate bone marrow reserve (absolute granulocyte count ≥2000/ml, platelet count ≥100000/ml); and adequate renal, hepatic, and cardiac function; ECOG performance status of 2 or less.

Patients were excluded from RSSH if they had any of the following: significant cardiopulmonary disease or contraindications for prolonged Trendelenburg position; prior pelvic or abdominal radiotherapy; severe hip disease limiting dorsolithotomy position. Previous abdominal surgery did not disqualify patients from the robotic approach.

Informed consent, including clinical evaluation and robotic single-port surgery, was obtained from all patients in accordance with local and international legislation (Declaration of Helsinki). All cases were performed on Vinci Single-Site® surgical system (Intuitive Surgical Inc®, 1266 Kifer Road, Building 101 Sunnyvale, CA) and the surgical team consisted of the primary surgeon (E.V.), bedside assistant and a robotics-dedicated scrub technician and circulating nurse.

Clinical patient characteristics included age, body mass index (BMI), clinical stage according to FIGO, and tumor grade. Moreover, status of the surgical margins and length of hospitalization, were evaluated. The time of the operation was subdivided into: (1) docking time, the time from the moment of port placement until the second robotic arm is mounted to the corresponding cannula; (2) console time, the actual surgical time, measured from the moment the surgeon starts maneuvering the surgical instruments until he orders their retrieval; and (3) operation time, the total skin-to-skin time. Intraoperative parameters included complications, blood loss, and hemoglobin levels before and 24 hours post-surgery. Blood transfusions were administered if hemoglobin was ≤ 7 g/L. Postoperative complications were assessed both short-term (within 30 days) and long-term (beyond 30 days), focusing on surgical, cardiac, pulmonary, and other events.

Pain was evaluated using a numeric rating scale (NRS) from 0 (no pain) to 10 (agonizing pain) at several intervals post-surgery. Analgesics included continuous infusion of tramadol and ketorolac for the first 24 hours, with paracetamol available on request. The cosmetic results of the umbilical scar were assessed by both patients and surgeons on days 1 and 30 post-surgery, with satisfaction rated from 0 (poor) to 10 (excellent).

Surgical procedure:

After indocyanine intracervical injection we used swabs to buffer the vagina. The cervix was closed and no uterus manipulator devices were used, but the cervix was closed with a modified tenaculum called "simple nebs arising incision landmark" (SNAIL®).

The first step started with an initial access, with an 2,5 cm long incision made over the lower rim of the umbilicus down to the level of the fascia, which was opened along the longitudinal axis of the body.

The leading edge of the folded port was inserted into the incision with a downward motion while countertraction was provided by retractors within the incision. An Intuitive Access Port of small size is placed into the incision and pneumoperitoneum is established by insufflating the abdomen to a pressure of 12 mm Hg. Patients were then placed in the steep Trendelenburg, low-lithotomy position, and the Da Vinci SP robot was docked laterally to the patients on the left side.

The Intuitive Access Port has four different channel port: in the superior channel was inserted a three-dimension 8.5mm optics,in channel number 1 was inserted a Cadiere Forceps, in channel number 2 a Maryland Bipolar and in channel number 3 a Monopolar Scissors (MCS). All instruments, including the camera, are articulating.

A careful inspection of the entire abdominal cavity was performed to identify any suspicious peritoneal lesion that would exclude the patient from having the procedure completed by robotic SP: the inspection is performed by inserting only the optics into the port. Afterward, all other instruments are introduced, and we proceeded with the surgical operation. After resection of the round ligament and an incision of the retroperitoneum over the course of the iliac external vessels, the ureter was visualized, a window was opened between the ovarian pedicle above and the ureter below, and ovarian pedicles were coagulated with Maryland Bipolar and resected with MCS. Next, we developed the retroperitoneal spaces (paravesical space, Lasko fossa, medial pararectal fossa, or Okabayashi pararectal space) from the right side to the left, identified the sentinel node on each side using Firefly, and removed it. Afterward, a type A hysterectomy was performed as described by Querleu and Morrow and uterine vessels were coagulated with Maryland Bipolar and resected with MCS. Colpotomy was performed with the MCS. The uterus and the adnexa were extracted through the vagina and sent for frozen section analysis. The vaginal vault was closed with a continuous suture using V-Loc and a needle driver instead of MCS. Finally, according to the frozen section results, we performed the systematic lymphadenectomy: following the guidelines, we performed lymphadenectomy only in patients with intermediate or high risk.

The arrangement of the instruments is the same as for hysterectomy. Lymphadenectomy is divided in three steps:

* First step: the surgeon prepares the medial limit of the lymphadenectomy starting from the common iliac artery following the hypogastric artery and the obliterated umbilical artery.
* Second step: the lateral limit is prepared by detaching pelvic vessels from the muscular surface of the pelvis
* Third step: the periadventitial plate of the common iliac artery and the external iliac artery is incised in a centrifugal direction and the lymph nodes are removed "en bloc" up to the obturator nerve. The lymph nodes are insert in an endobag and removed through the vaginal canal before the vagina is sutured.

ELIGIBILITY:
Inclusion Criteria: Patients with clinically confirmed endometrioid endometrial cancer, FIGO stage IA-IB.

-

Exclusion Criteria: significant cardiopulmonary disease or contraindications for prolonged Trendelenburg position; prior pelvic or abdominal radiotherapy; severe hip disease limiting dorsolithotomy position

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-06-26 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Operative Time | during the intervention/procedure/surgery
  duration of the hysterectomy, measured in minutes
Docking Time | during the intervention/procedure/surgery
  Duration of the davinci SP docking, measured in minutes
Console Time | during the intervention/procedure/surgery
  Time spent by the surgeon in the console during the surgical operation, measured in minutes
Blood loss | during the intervention/procedure/surgery
  Blood loss during the surgery, measured in ml
Change in hemoglobin | immediately after the intervention/procedure/surgery
  Change in hemoglobin after the surgery, measured in g/dl

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS regina elena cancer istitute, Rome, rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Background] Barletta F, Corrado G, Vizza E. Laparoscopic radical hysterectomy with the use of SNAIL Tenaculum™. A simplified uterine manipulator for the management of early cervical cancer
- [Background] Pecorelli S. Revised FIGO staging for carcinoma of the vulva, cervix, and endometrium. Int J Gynaecol Obstet. 2009 May;105(2):103-4. doi: 10.1016/j.ijgo.2009.02.012. No abstract available. PMID 19367689
- [Background] Nguyen TT, Basilius J, Ali SN, Dobbs RW, Lee DI. Single-Port Robotic Applications in Urology. J Endourol. 2023 Jun;37(6):688-699. doi: 10.1089/end.2022.0600. Epub 2023 May 15. PMID 37029799
- [Background] Jung JM, Kim YI, Yoon YS, Yang S, Kim MH, Lee JL, Kim CW, Park IJ, Lim SB, Yu CS. Short-term outcomes of da Vinci SP versus Xi for colon cancer surgery: a propensity-score matching analysis of multicenter cohorts. J Robot Surg. 2023 Dec;17(6):2911-2917. doi: 10.1007/s11701-023-01727-3. Epub 2023 Oct 11. PMID 37821761
- [Background] Arcieri, P. Romeo, G Vizzielli, S. Restaino, L. Driul, G. Stabile, R. Granese, S. Cianci, A. Ercoli. (2023). Robotic Single-Port da Vinci Surgical System (SP1098) in Gynecologic Surgery: A Systematic Review of Literature. Clinical and Experimental Obstetrics and Gynecology.
- [Background] Cianci S, Rosati A, Rumolo V, Gueli Alletti S, Gallotta V, Turco LC, Corrado G, Vizzielli G, Fagotti A, Fanfani F, Scambia G, Uccella S. Robotic Single-Port Platform in General, Urologic, and Gynecologic Surgeries: A Systematic Review of the Literature and Meta-analysis. World J Surg. 2019 Oct;43(10):2401-2419. doi: 10.1007/s00268-019-05049-0. PMID 31187247
- [Background] Corrado G, Calagna G, Cutillo G, Insinga S, Mancini E, Baiocco E, Zampa A, Bufalo A, Perino A, Vizza E. The Patient and Observer Scar Assessment Scale to Evaluate the Cosmetic Outcomes of the Robotic Single-Site Hysterectomy in Endometrial Cancer. Int J Gynecol Cancer. 2018 Jan;28(1):194-199. doi: 10.1097/IGC.0000000000001130. PMID 29040189
- [Background] Bianco FM, Dreifuss NH, Chang B, Schlottmann F, Cubisino A, Mangano A, Pavelko Y, Masrur MA, Giulianotti PC. Robotic single-port surgery: Preliminary experience in general surgery. Int J Med Robot. 2022 Dec;18(6):e2453. doi: 10.1002/rcs.2453. Epub 2022 Aug 19. PMID 35962708
- [Derived] Vizza R, Corrado G, Mancini E, Baiocco E, Russo M, Vincenzoni C, Bruno V, Falconer H, Vizza E. Feasibility, safety, and efficacy of robotic single-port hysterectomy (R-SPH) using the da Vinci SP system in low-risk endometrial cancer: a pilot study. Minim Invasive Ther Allied Technol. 2025 Dec;34(6):433-440. doi: 10.1080/13645706.2025.2538764. Epub 2025 Aug 11. PMID 40788153